CLINICAL TRIAL: NCT05093894
Title: A Prospective, Multicenter Randomized Study of Microlyte - AG Bioresorbable Matrix in the Prevention of Surgical Site Infection After Open Ventral Hernia Repair
Brief Title: Microlyte in Prevention of SSI After Open Ventral Hernia Repair
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: PI decided not to continue study due to no funding.
Sponsor: Prisma Health-Upstate (Other)
Collaborators: Wake Forest University Health Sciences (Other); Kendall Healthcare Group, Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pro00115720
Record Dates: First submitted 2021-10-13; First posted 2021-10-26 (Actual); Last update posted 2022-10-10 (Actual); Status verified 2022-10

CONDITIONS: Ventral Hernia
MeSH Terms: conditions — Hernia, Ventral

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Group 1: Microlyte will be cut into strips and placed on the surgical incision (Active Comparator): Microlyte will be cut into strips and placed on the surgical incision
  Interventions: Device: Group 1
- Group 2: Nothing will be placed on the surgical incision (No Intervention): Nothing will be placed on the surgical incision

INTERVENTIONS:
Device: Group 1 — Microlyte will be cut into strips and placed on the subcutaneous space
  Arms: Group 1: Microlyte will be cut into strips and placed on the surgical incision

SUMMARY:
Participants who are scheduled to have open ventral hernia repair (OVHR) will be asked to take part in this study.

The purpose of this study is to find out if placing Microlyte (which is a dissolvable sheet coated in silver) on the surgical incision is better than placing nothing on the surgical incision when it comes to decreasing the chance of surgical site infections.

The study device has been cleared by the Food and Drug Administration (FDA) for use on surgical incisions.

A total of 280 participants will be included in the study.

Participation will last for about 90 days.

DETAILED DESCRIPTION:
The aim of our study is to assess the impact of Microlyte-AG® (Imbed Biosciences, Fitchburg, WI), a silver-coated bioabsorbable matrix, on surgical site infection (SSI) on patients undergoing clean open ventral hernia repair (OVHR) at Carolinas Medical Center/Atrium Health (Charlotte, NC), Prisma Health-Upstate (Greenville, SC), and Mission Health/HCA Healthcare (Asheville, NC).

Those who agree to participate in the study will undergo the following:

Information will be collected, including demographics, past medical and surgical history, and hospital outcomes.

On the day of surgery, participants will be "randomized" into one of the study groups listed below.

* Group 1: The study device will be cut into strips and placed in the surgical incision
* Group 2: Nothing will be placed in the surgical incision

For both groups, the surgical incision will then be closed with absorbable sutures, which is the usual treatment.

Participants will be seen by the study doctor 30 and 90 days after surgery for a checkup. At the 30-day visit, participants will have a physical examination, and the study doctor will check to see if any complications have happened since the last visit. The 90-day follow-up visit can be done in person or over the telephone and will be done to check and see if there have been any problems with the healing of the surgical incision.

ELIGIBILITY:
Inclusion Criteria:

* Men and women over 18 years of age
* Patients undergoing open hernia repair with retromuscular or preperitoneal placement of polypropylene mesh in clean (Class I) operative fields, and who are candidates for complete skin closure
* Capable and willing to attend the scheduled postoperative visits
* Signed ICF for study enrollment

Exclusion Criteria:

* Prisoners
* Minimally invasive repairs (laparoscopy, robotics)
* CDC Wound Class II-IV
* Irrigation of the wound or peritoneal cavity with antibiotic or antimicrobial fluid
* Inability to completely close the midline fascia
* Mesh placed as a bridge, onlay, or intraperitoneal position to the fascia
* Skin left open or packed at the time of the index operation
* Use of wound wicks at the time of the index operation
* Use of an investigational product within the preceding 60 days
* Allergy to silver

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-12-14 (Actual); Primary Completion 2022-10-06 (Actual); Study Completion 2022-10-06 (Actual)

PRIMARY OUTCOMES:
Rate of SSI following clean OVHR with and without Microlyte. | 90 days
  SSI, which is the primary outcome that will be measured for the study will be as an infection of the skin or subcutaneous tissues as clinically determined by the physician caring for the patient

SECONDARY OUTCOMES:
Rate of other wound complications, including superficial wound breakdown, seroma formation, and mesh infection, with/without Microlyte. | 90 days
  Other wound complications will be defined based on a combination of clinical assessment and review of postoperative notes and imaging
Rate of short-term readmissions with and without Microlyte | 30-days
  Short-term readmissions

CONTACTS AND LOCATIONS:
Overall Officials: Alfredo M Carbonell, DO, Principal Investigator — Prisma Health
Locations (3):
- United States (3):
  - Mission Hospital/HCA Healthcare, Asheville, North Carolina
  - Carolinas Medical Center/Atrium Health, Charlotte, North Carolina
  - Prisma Health, Greenville, South Carolina

IPD SHARING:
Plan to Share IPD: No